CLINICAL TRIAL: NCT00274872
Title: Phase II-III Study of an Optimized LV-5FU-Oxaliplatin Strategy in Metastatic Colorectal Cancer. Optimox2 Study. C02-2
Brief Title: Combination Chemotherapy in Treating Patients With Metastatic Colorectal Cancer That Cannot Be Removed By Surgery
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000453890; GERCOR-OPTIMOX2; GERCOR-OPTIMOX2-2003; GERCOR-OPTIMOX2-C02-2; EU-20566; SANOFI-GERCOR-OPTIMOX2
Record Dates: First submitted 2006-01-10; First posted 2006-01-11 (Estimated); Last update posted 2010-02-01 (Estimated); Status verified 2007-05

CONDITIONS: Colorectal Cancer
Keywords: recurrent rectal cancer; stage IV rectal cancer; recurrent colon cancer; stage IV colon cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms; Colonic Neoplasms | interventions — Fluorouracil; Leucovorin; Oxaliplatin

INTERVENTIONS:
Drug: fluorouracil
Drug: leucovorin calcium
Drug: oxaliplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as oxaliplatin, leucovorin, and fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells. It is not yet known which combination chemotherapy regimen is more effective in treating colorectal cancer.

PURPOSE: This randomized phase II/III trial is studying two combination chemotherapy regimens to compare how well they work in treating patients with metastatic colorectal cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare progression-free survival of patients with inoperable metastatic colorectal cancer treated with oxaliplatin, leucovorin calcium, and fluorouracil with vs without maintenance leucovorin calcium and fluorouracil.
* Demonstrate that time of disease control (TDC) can be increased by 15% at 9 months and that maintenance therapy can be avoided.

Secondary

* Compare the overall survival and response rate in patients treated with these regimens.
* Compare the salvage surgery rate in patients treated with these regimens.
* Compare the tolerability of these regimens in these patients.
* Compare the quality of life in patients treated with these regimens.
* Compare the duration of chemotherapy-free intervals in patients treated with these regimens.
* Compare the pharmacoeconomy and pharmacogenetics of these regimens in these patients.

OUTLINE: This is a randomized, controlled, open-label, multicenter study. Patients are stratified according to participating center, performance status (0-1 vs 2), number of metastatic sites (1 vs > 1), age (18-50 years vs 51-75 years vs 76-80 years), adjuvant chemotherapy, and baseline alkaline phosphatase (≤ 3 times upper limit of normal [ULN] vs > 3 times ULN). Patients are randomized to 1 of 2 treatment arms.

Arm I

* FOLFOX chemotherapy: Patients receive oxaliplatin IV over 2 hours and leucovorin calcium IV over 2 hours on day 1 and fluorouracil IV continuously over 46 hours on days 1 and 2. Treatment repeats every 14 days for 6 courses in the absence of disease progression or unacceptable toxicity. Patients then proceed to maintenance chemotherapy.
* Maintenance chemotherapy: Patients receive leucovorin calcium IV over 2 hours on day 1 and fluorouracil IV continuously over 46 hours on days 1 and 2. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.

Patients with disease progression on maintenance chemotherapy receive 6 additional courses of FOLFOX as above. Patients with continued disease progression while receiving the additional courses of FOLFOX proceed to irinotecan-based chemotherapy off study.

Arm II

* FOLFOX chemotherapy: Patients receive 6 courses of FOLFOX as in arm I. Patients with disease progression on FOLFOX receive 6 additional courses of FOLFOX. Patients with continued disease progression while receiving the additional courses of FOLFOX proceed to irinotecan-based chemotherapy off study.

In both arms, patients with stable or responding disease may undergo surgical resection after completion of the initial 6 courses of FOLFOX.

Quality of life is assessed at baseline, after courses 4 and 6, and then every 2-3 months thereafter.

After completion of study treatment, patients are followed at 1 month and then every 3 months thereafter.

PROJECTED ACCRUAL: A total of 600 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven adenocarcinoma of the colon or rectum

  * Metastatic disease

    * No metastases involving only the bone
* Inoperable disease (i.e., not suitable for complete surgical resection)
* Measurable or evaluable disease

  * Measurable disease defined as ≥ 1 unidimensionally measurable lesion ≥ 20 mm by conventional CT scan OR ≥ 10 mm by spiral CT scan
* No symptomatic ascites or pleural effusion that has not been evacuated
* No CNS metastasis

PATIENT CHARACTERISTICS:

* WHO OR ECOG performance status 0-2
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelets ≥ 100,000/mm^3
* Creatinine < 3 times upper limit of normal (ULN)
* Alkaline phosphatase < 5 times ULN
* No peripheral neuropathy ≥ grade 1
* No total or partial bowel obstruction
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No uncontrolled hypercalcemia
* No other concurrent or prior malignancy, except adequately treated carcinoma in situ of the uterine cervix or basal or squamous cell carcinoma of the skin or cancer in complete remission for ≥ 5 years
* No uncontrolled congestive heart failure
* No angina pectoris
* No hypertension
* No arrhythmias
* No history of significant neurologic or psychiatric disorders
* No active infection
* No other serious nonmalignant disease

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy and/or immunotherapy for metastatic disease
* Prior adjuvant chemotherapy allowed provided progression-free interval after completion of adjuvant chemotherapy is > 6 months
* No other concurrent anticancer treatment
* No participation in another clinical trial with any investigational drug within 30 days prior to randomization
* No other concurrent investigational treatment
* No concurrent radiotherapy
* No concurrent cold cap for prevention of alopecia or iced mouth rinses for prevention of stomatitis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2004-01

PRIMARY OUTCOMES:
Overall survival
Time to disease control
Response as measured by RECIST criteria
Toxicity
Quality of life as assessed by EUROQOL- 5 Dimensional Instrument or Functional Assessment of Cancer Therapy-Neurotoxicity module version 4.0 at baseline and periodically during study treatment
Pharmaco-economic evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Aimery de Gramont, MD, Study Chair — Hopital Saint Antoine
Locations (17):
- France (17):
  - Institut Sainte Catherine, Avignon
  - Hopital Duffaut, Avignon
  - Infirmerie Protestante, Caluire-et-Cuire
  - Hopital Drevon, Dijon
  - Centre Hospitalier de Dreux, Dreux
  - Hopital Louis Pasteur - Le Coudray, Le Coudray
  - Clinique Victor Hugo, Le Mans
  - Hopital Robert Boulin, Libourne
  - Clinique Saint Jean, Lyon
  - Intercommunal Hospital, Montfermeil
  - Hopital Europeen Georges Pompidou, Paris
  - Hopital Saint Antoine, Paris
  - Hopital Tenon, Paris
  - Polyclinique De Courlancy, Reims
  - C.H. Senlis, Senlis
  - Clinique des Jockeys, Senlis
  - Centre Medico-Chirurgical Foch, Suresnes

REFERENCES:
- [Result] Chibaudel B, Maindrault-Goebel F, Lledo G, Mineur L, Andre T, Bennamoun M, Mabro M, Artru P, Carola E, Flesch M, Dupuis O, Colin P, Larsen AK, Afchain P, Tournigand C, Louvet C, de Gramont A. Can chemotherapy be discontinued in unresectable metastatic colorectal cancer? The GERCOR OPTIMOX2 Study. J Clin Oncol. 2009 Dec 1;27(34):5727-33. doi: 10.1200/JCO.2009.23.4344. Epub 2009 Sep 28. PMID 19786657